CLINICAL TRIAL: NCT04585750
Title: A Phase 1/2 Open-label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of PC14586 in Patients With Locally Advanced or Metastatic Solid Tumors Harboring a TP53 Y220C Mutation (PYNNACLE)
Brief Title: The Evaluation of PC14586 in Patients With Advanced Solid Tumors Harboring a TP53 Y220C Mutation (PYNNACLE)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PMV Pharmaceuticals, Inc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMV-586-101; KEYNOTE-D79 (Registry Identifier: Merck, Sharp & Dohme, LLC); MK-3475-D79 (Registry Identifier: Merck, Sharp & Dohme, LLC)
Record Dates: First submitted 2020-10-01; First posted 2020-10-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; Advanced Malignant Neoplasm; Metastatic Cancer; Metastatic Solid Tumor; Lung Cancer; Ovarian Cancer; Endometrial Cancer; Prostate Cancer; Colorectal Cancer; Breast Cancer; Other Cancer; Locally Advanced; Head and Neck Cancer; Gall Bladder Cancer; Small Cell Lung Cancer; Small Cell Lung Cancer ( SCLC ); Small Cell Lung Carcinoma; NSCLC; NSCLC (Non-small Cell Lung Cancer); SCLC; Non-Small Cell Lung Carcinoma; Triple Negative Breast Cancer; TNBC; HER2+ Breast Cancer; Non-Small Cell Lung Cancer; ER/PR Positive Breast Cancer; HER2- Breast Cancer; HER2-positive Breast Cancer; HER2-negative Breast Cancer; ER/PR(+), Her2(-) Breast Cancer
Keywords: PC14586; p53; Y220C; Phase 1; Phase 1/2; PMV; PMV Pharma; p53 mutation; TP53; TP53 mutation; p53 mutant; p53 reactivator; pembrolizumab; Keytruda; combination; PD-1; PD-L1; anti-PD-1; Merck; MSD; IgG4; mAb; Phase 1b; NGS; Next Generation Sequencing; precision; Phase 2; Rezatapopt
MeSH Terms: conditions — Neoplasm Metastasis; Lung Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Head and Neck Neoplasms; Gallbladder Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: During Phase 2 Monotherapy, 2000mg QD of PC14586 (INN: rezatapopt) will be assigned to all participants. Participants will be assigned to one of five cohorts: ovarian cancer, lung cancer, breast cancer, endometrial cancer, or other solid tumors. Enrollment ongoing.
  During Phase 1 Monotherapy (Dose Escalation), participants will be assigned a dose level using an accelerated titration design in the initial dose cohorts, followed by a modified toxicity probability interval (mTPI) design in subsequent dose cohorts. Enrollment closed.
  During Part 1 of the Ph 1b Combination Therapy, patients will be assigned a dose level using mTPI design. A recommended rezatapopt Phase 2 Dose (RP2D) when administered in combination with pembrolizumab will be selected at the end of Phase 1b Part 1, and the RP2D will be assigned to all participants in Part 2. Enrollment closed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Phase 1 Monotherapy Dose Escalation (Experimental): Multiple dose levels of daily oral rezatapopt will be evaluated in an escalating manner, to determine the maximum tolerated dose and to ensure sufficient safety experience, pharmacokinetic information, and early evidence of clinical activity of rezatapopt to recommend a Phase 2 dose (RP2D).
  Interventions: Drug: rezatapopt
- Phase 1b Combination Therapy Dose Escalation, Part 1 (Experimental): Multiple dose levels of daily oral rezatapopt in combination with a stable dose of pembrolizumab (200 mg IV q3 weeks) will be evaluated in an escalating manner, to determine the maximum tolerated dose and to ensure sufficient safety experience, pharmacokinetic information, and early evidence of clinical activity of PC14586 to recommend a Phase 2 dose (RP2D) of rezatapopt when administered in combination with pembrolizumab.
  Interventions: Drug: rezatapopt; Drug: pembrolizumab
- Phase 1b Combination Therapy Dose Expansion, PD(L)-1 naive patients (Experimental): Additional (expansion of) participants will enroll at the RP2D of daily oral PC14586 (INN: rezatapopt) when administered in combination with pembrolizumab (200 mg IV q3 weeks) for continued evaluation. Participants will have advanced solid tumors harboring a p53 Y220C mutation and are PD(L)-1 naive patients.
  Interventions: Drug: rezatapopt; Drug: pembrolizumab
- Phase 1b Combination Therapy Dose Expansion, PD(L)-1 relapsed/refractory patients (Experimental): Additional (expansion of) participants will enroll at the RP2D of daily oral rezatapopt when administered in combination with pembrolizumab (200 mg IV q3 weeks) for continued evaluation. Participants will have advanced solid tumors harboring a p53 Y220C mutation and are PD(L)-1 relapsed/refractory patients.
  Interventions: Drug: rezatapopt; Drug: pembrolizumab
- Phase 2 Monotherapy Dose Expansion, Ovarian Cancer Cohort (Experimental): Additional (expansion of) participants will dose with 2000 mg daily oral PC14586 (INN: rezatapopt) with food for continued evaluation. Ovarian Cancer Cohort participants will have locally advanced or metastatic ovarian cancer harboring a TP53 Y220C mutation who meet all eligibility criteria and have measurable disease per RECIST 1.1.
  Interventions: Drug: rezatapopt
- Phase 2 Monotherapy Dose Expansion, Lung Cancer Cohort (Experimental): Additional (expansion of) participants will dose with 2000 mg daily oral PC14586 (INN: rezatapopt) with food for continued evaluation. Lung Cancer Cohort participants will have locally advanced or metastatic lung cancer harboring a TP53 Y220C mutation who meet all eligibility criteria and have measurable disease per RECIST 1.1.
  Interventions: Drug: rezatapopt
- Phase 2 Monotherapy Dose Expansion, Breast Cancer Cohort (Experimental): Additional (expansion of) participants will dose with 2000 mg daily oral PC14586 (INN: rezatapopt) with food for continued evaluation. Breast Cancer Cohort participants will have locally advanced or metastatic breast cancer harboring a TP53 Y220C mutation who meet all eligibility criteria and have measurable disease per RECIST 1.1.
  Interventions: Drug: rezatapopt
- Phase 2 Monotherapy Dose Expansion, Endometrial Cancer Cohort (Experimental): Additional (expansion of) participants will dose with 2000 mg daily oral PC14586 (INN: rezatapopt) with food for continued evaluation. Endometrial Cancer Cohort participants will have locally advanced or metastatic endometrial cancer harboring a TP53 Y220C mutation who meet all eligibility criteria and have measurable disease per RECIST 1.1.
  Interventions: Drug: rezatapopt
- Phase 2 Monotherapy Dose Expansion, Other Solid Tumors Cohort (Experimental): Additional (expansion of) participants will dose with 2000 mg daily oral PC14586 (INN: rezatapopt) with food for continued evaluation. Other Solid Tumors Cohort participants will have locally advanced or metastatic solid tumors harboring a TP53 Y220C mutation who meet all eligibility criteria and have measurable disease per RECIST 1.1.
  Interventions: Drug: rezatapopt

INTERVENTIONS:
Drug: rezatapopt — First-in-class, oral, small molecule p53 reactivator selective for the TP53 Y220C mutation.
  Other Names: PC14586
Drug: pembrolizumab — Participants receive pembrolizumab 200 mg by intravenous (IV) infusion over 30 minutes.
  Other Names: KEYTRUDA®; MK-3475; KEYNOTE-D79; MK-3475-D79
  Arms: Phase 1b Combination Therapy Dose Escalation, Part 1; Phase 1b Combination Therapy Dose Expansion, PD(L)-1 naive patients; Phase 1b Combination Therapy Dose Expansion, PD(L)-1 relapsed/refractory patients

SUMMARY:
The Phase 2 monotherapy portion of this study is currently enrolling and will evaluate the efficacy and safety of PC14586 (INN rezatapopt) in participants with locally advanced or metastatic solid tumors harboring a TP53 Y220C mutation. The Phase 1 portion of the study will assess the safety, tolerability and preliminary efficacy of multiple dose levels of rezatapopt as monotherapy and in Phase 1b in combination with pembrolizumab.

DETAILED DESCRIPTION:
Rezatapopt is a first-in-class, oral, small molecule p53 reactivator that is selective for the TP53 Y220C mutation.

The primary objective of Phase 2 Monotherapy is to evaluate the efficacy of rezatapopt at the Recommended Phase 2 Dose (RP2D) including the Overall Response Rate (ORR) in the Ovarian Cancer Cohort and the ORR across all cohorts as determined by blinded independent central review. Secondary objectives of Phase 2 are to characterize the safety, pharmacokinetic (PK) properties, quality of life, and other efficacy measures of PC14586 rezatapopt at the RP2D. Enrollment is open for the Phase 2 Monotherapy portion of the study.

The primary objective of Phase 1 Monotherapy is to establish the maximum tolerated dose (MTD) and RP2D of rezatapopt. Secondary objectives are to characterize the PK properties, safety and tolerability, and to assess preliminary efficacy including ORR. Enrollment into Phase 1 Monotherapy is complete.

The primary objective of Phase 1b Combination Therapy is to establish the MTD/RP2D of rezatapopt when administered in combination with pembrolizumab. Secondary objectives of Phase 1b Combination Therapy are to characterize PK, safety and tolerability, and to assess preliminary efficacy of rezatapopt when administered in combination with pembrolizumab, including ORR. Enrollment into Phase 1b Combination Therapy is complete.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age or 12 to 17 years of age after Safety Review Committee approval.
* Locally advanced or metastatic solid malignancy with a TP53 Y220C mutation
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Previously treated with one or more lines of anticancer therapy and progressive disease
* Adequate organ function
* Measurable disease per RECIST v1.1 (Phase 2)

Additional Criteria for Inclusion in Phase 1b (rezatapopt) + pembrolizumab combination)

* Anti-PD-1/PD-L1 naive or must have progressed on treatment
* Measurable disease

Exclusion Criteria:

* Anti-cancer therapy within 21 days (or 5 half-lives) of receiving the study drug
* Radiotherapy within 14 days of receiving the study drug
* Primary CNS tumor
* History of leptomeningeal disease or spinal cord compression
* Brain metastases, unless neurologically stable and do not require steroids to treat associated neurological symptoms
* Stroke or transient ischemic attack within 6 months prior to screening
* Heart conditions such as unstable angina within 6 months prior to screening, uncontrolled hypertension, a heart attack within 6 months prior to screening, congestive heart failure, prolongation of QT interval, or other rhythm abnormalities
* Strong CYP3A4 inducers and strong CYP2C9 inhibitors/inducers within 14 days of first dose of rezatapopt
* History of gastrointestinal (GI) disease that may interfere with absorption of study drug or patients unable to take oral medication
* History of prior organ transplant
* Known, active malignancy, except for treated cervical intraepithelial neoplasia, or non-melanoma skin cancer
* Known, active uncontrolled Hepatitis B, Hepatitis C, or human immunodeficiency virus infection

Additional Criteria for Exclusion from Phase 2 (rezatapopt monotherapy)

* Known KRAS mutation, defined as a single nucleotide variant (SNV) (Phase 2)

Additional Criteria for Exclusion from Phase 1b (rezatapopt) + pembrolizumab combination)

* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor and discontinued from that treatment due to a Grade 3 or higher immune-related AE (irAE)
* Received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention
* Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy within 7 days prior to the first dose of study drug
* Hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients
* Active autoimmune disease that has required systemic treatment in past 2 years
* History of radiation pneumonitis
* History of (non-infectious) or active pneumonitis / interstitial lung disease that required steroids
* Active infection requiring systemic therapy
* Known history of HIV infection
* Has previously received rezatapopt

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Monotherapy (Dose Escalation): Determine the number and type of adverse events to characterize the safety of rezatapopt | 40 months
  Number of participants with treatment related adverse events
Phase 1 Monotherapy (Dose Escalation): Establish the Recommended Phase 2 Dose (RP2D) | 30 months
  RP2D will be determined using available safety and pharmacokinetics and pharmacodynamics data
Phase 1 Monotherapy (Dose Escalation): Establish the maximum tolerated dose (MTD) (Phase 1) | The first 28 days of treatment (Cycle 1) per patient
  Incidence of dose limiting toxicities (DLTs) during the first 28 days of treatment with rezatapopt
Phase 1b Combination Therapy (Part 1: Dose Escalation): Determine the number and type of adverse events to characterize the safety of rezatapopt when administered in combination with pembrolizumab | 18 months for treatment arm
  Number of participants with treatment related adverse events
Phase 1b Combination Therapy (Part 1: Dose Escalation): Establish the maximum tolerated dose (MTD) of rezatapopt when administered in combination with pembrolizumab | The first 28 days of combination treatment arm (starting on Day -7) per patient
  Incidence of dose limiting toxicities (DLTs) during the first 28 days of treatment with rezatapopt
Phase 1b Combination Therapy (Part 1: Dose Escalation): Establish the Recommended Phase 2 Dose (RP2D) of rezatapopt when administered in combination with pembrolizumab | 18 months
  RP2D will be determined using available safety and pharmacokinetics and pharmacodynamics data
Phase 1b Combination Therapy (Part 2: Dose Expansion): Determine the number and type of adverse events to characterize the safety of rezatapopt when administered in combination with pembrolizumab | 12 months for treatment arm
  Number of participants with treatment related adverse events
Phase 2 Monotherapy (Dose Expansion): Response rate assessment to evaluate the clinical activity / efficacy of rezatapopt | 34 months
  Overall response rate in accordance with Response Evaluation Criteria (RECIST) v.1.1 as assessed by independent review across all cohorts
Phase 2 Monotherapy (Dose Expansion): Response rate assessment to evaluate the clinical activity / efficacy of rezatapopt in ovarian cancer patients | 34 months
  Overall response rate in accordance with Response Evaluation Criteria (RECIST) v.1.1 as assessed by independent review in the ovarian cancer cohort

SECONDARY OUTCOMES:
Phase 1 Monotherapy: PK profile of rezatapopt - Peak concentration (Cmax) | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 1 Monotherapy: PK profile of rezatapopt - Time of peak concentration (Tmax) | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 1 Monotherapy: PK profile of rezatapopt - Area under the plasma concentration-time curve from time zero to time of last sampling timepoint (AUC0-t) | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 1 Monotherapy: PK profile of rezatapopt - Area under the plasma concentration-time curve in one dosing interval (AUCtau) | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 1 Monotherapy: PK profile of rezatapopt - Trough observed concentrations (Ctrough/Ctau) | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 1 Monotherapy: Blood plasma assessment to describe the concentration of PC14586 and metabolites when rezatapopt is administered orally. | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Blood plasma concentration
Phase 1 Monotherapy (Dose Escalation): Overall Response Rate per RECIST v1.1 or PCWG3 modified RECIST v1.1 | 41 months for study (end of Phase 1)
  Evaluation of preliminary anti-tumor activity of rezatapopt as a single agent
Phase 1 Monotherapy (Dose Escalation): Time to Response per RECIST v1.1 or PCWG3 modified RECIST v1.1 | 41 months for study (end of Phase 1)
  Evaluation of preliminary anti-tumor activity of rezatapopt as a single agent
Phase 1 Monotherapy (Dose Escalation): Duration of Response per RECIST v1.1 or PCWG3 modified RECIST v1.1 | 41 months for study (end of Phase 1)
  Evaluation of preliminary anti-tumor activity of rezatapopt as a single agent
Phase 1 Monotherapy (Dose Escalation): Disease Control Rate per RECIST v1.1 or PCWG3 modified RECIST v1.1 | 41 months for study (end of Phase 1)
  Evaluation of preliminary anti-tumor activity of rezatapopt as a single agent
Phase 1 Monotherapy (Dose Escalation): Progression Free Survival per RECIST v1.1 or PCWG3 modified RECIST v1.1 | 41 months for study (end of Phase 1)
  Evaluation of preliminary anti-tumor activity of rezatapopt as a single agent
Phase 1 Monotherapy (Dose Escalation): Overall Survival | 41 months for study (end of Phase 1)
  Evaluation of preliminary anti-tumor activity of rezatapopt as a single agent
Phase 1b Combination Therapy: PK profile of rezatapopt in combination with pembrolizumab - Peak concentration (Cmax) | Approximately 12 months per patient (30 months for treatment arm)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 1b Combination Therapy: PK profile of rezatapopt in combination with pembrolizumab - Time of peak concentration (Tmax) | Approximately 12 months per patient (30 months for treatment arm)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 1b Combination Therapy: PK profile of rezatapopt in combination with pembrolizumab - Area under the plasma concentration-time curve from time zero to time of last sampling timepoint (AUC0-t) | Approximately 12 months per patient (30 months for treatment arm)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 1b Combination Therapy: PK profile of rezatapopt in combination with pembrolizumab - Area under the plasma concentration-time curve in one dosing interval (AUCtau) | Approximately 12 months per patient (30 months for treatment arm)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 1b Combination Therapy: PK profile of rezatapopt in combination with pembrolizumab - Trough observed concentrations (Ctrough/Ctau) | Approximately 12 months per patient (30 months for treatment arm)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 1b Combination Therapy: Blood plasma assessment to describe the concentration of rezatapopt and metabolites when rezatapopt is administered orally in combination with pembrolizumab. | Approximately 12 months per patient (30 months for treatment arm)
  Blood plasma concentration
Phase 1b Combination Therapy: Overall Response Rate per RECIST v1.1, iRECIST, or PCWG3 as assessed by Investigator and as assessed by independent review | 30 months for study (end of Phase 1b)
  Evaluation of anti-tumor activity of rezatapopt in combination with pembrolizumab
Phase 1b Combination Therapy: Time to Response per RECIST v1.1, iRECIST, or PCWG3 as assessed by Investigator and as assessed by independent review | 30 months for study (end of Phase 1b)
  Evaluation of anti-tumor activity of rezatapopt in combination with pembrolizumab
Phase 1b Combination Therapy: Duration of Response per RECIST v1.1, iRECIST, or PCWG3 as assessed by Investigator and as assessed by independent review | 30 months for study (end of Phase 1b)
  Evaluation of anti-tumor activity of rezatapopt in combination with pembrolizumab
Phase 1b Combination Therapy: Disease Control Rate per RECIST v1.1, iRECIST, or PCWG3 as assessed by Investigator and as assessed by independent review | 30 months for study (end of Phase 1b)
  Evaluation of anti-tumor activity of rezatapopt in combination with pembrolizumab
Phase 1b Combination Therapy: Overall Survival | 30 months for study (end of Phase 1b)
  Evaluation of anti-tumor activity of rezatapopt in combination with pembrolizumab
Phase 1b Combination Therapy: Determine the number and type of adverse events to characterize the safety of rezatapopt | 30 months for study (end of Phase 1b)
  Number of participants with treatment related adverse events
Phase 1b Combination Therapy: Progression Free Survival per RECIST v1.1, iRECIST, or PCWG3 as assessed by Investigator and as assessed by independent review | 30 months for study (end of Phase 1b)
  Evaluation of anti-tumor activity of rezatapopt in combination with pembrolizumab
Phase 2 Monotherapy: PK profile of rezatapopt - Time of peak concentration (Tmax) | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 2 Monotherapy: PK profile of rezatapopt - Peak concentration (Cmax) | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 2 Monotherapy: PK profile of rezatapopt - Area under the plasma concentration-time curve from time zero to time of last sampling timepoint (AUC0-t) | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 2 Monotherapy: PK profile of rezatapopt - Area under the plasma concentration-time curve in one dosing interval (AUCtau) | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 2 Monotherapy: PK profile of rezatapopt - Trough observed concentrations (Ctrough/Ctau) | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt
Phase 2 Monotherapy: Blood plasma assessment to describe the concentration of rezatapopt and metabolites when rezatapopt is administered orally. | Approximately 12 months per patient (75 months for Phase 1 and Phase 2)
  Blood plasma concentration
Phase 2 Monotherapy (Dose Expansion): Determine the number and type of adverse events to characterize the safety of rezatapopt | 34 months for study (end of Phase 2)
  Number of participants with treatment related adverse events
Phase 2 Monotherapy (Dose Expansion): Overall Response Rate across all cohorts per RECIST v1.1 as assessed by Investigator | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Overall Response Rate in ovarian cancer cohort per RECIST v1.1 as assessed by Investigator | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Time to Response in ovarian cancer cohort per RECIST v1.1 as assessed by Investigator and as assessed by independent review | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Time to Response across all cohorts per RECIST v1.1 as assessed by Investigator and as assessed by independent review | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Duration of Response in ovarian cancer cohort per RECIST v1.1 as assessed by Investigator and as assessed by independent review | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Duration of Response across all cohorts per RECIST v1.1 as assessed by Investigator and as assessed by independent review | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Disease Control Rate in ovarian cancer cohort per RECIST v1.1 as assessed by Investigator and as assessed by independent review | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Disease Control Rate across all cohorts per RECIST v1.1 as assessed by Investigator and as assessed by independent review | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Progression Free Survival in ovarian cancer cohort per RECIST v1.1 as assessed by Investigator and as assessed by independent review | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Progression Free Survival across all cohorts per RECIST v1.1 as assessed by Investigator and as assessed by independent review | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Overall Survival in ovarian cancer cohort | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Overall Survival across all cohorts | 34 months for study (end of Phase 2)
  Evaluation of anti-tumor activity of rezatapopt as a single agent
Phase 2 Monotherapy (Dose Expansion): Quality of life assessment | Evaluated at every visit. 34 months for treatment arm (end of Phase 2)
  Changes from baseline in quality of life as measured by a validated instrument, for participants 18 and older

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fellous, MD, Study Director — Sr. Vice President of Medical Affairs
Locations (75):
- United States (31):
  - University of California Irvine Chao Family Comprehensive Cancer Center, Irvine, California
  - University of San Diego Moores Cancer Center, La Jolla, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Advent Health, Orlando, Florida
  - Florida Cancer Specialists South, Port Charlotte, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering, New York, New York
  - Duke University, Durham, North Carolina
  - The Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - WellSpan York Cancer Center, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - New Experimental Therapeutics - NEXT Oncology, Austin, Texas
  - UTSW - Moody Outpatient Center - Parkland Health, Dallas, Texas
  - UT Southwest Simmons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - New Experimental Therapeutics of San Antonio - NEXT Oncology, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington, Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Australia (5):
  - Chris O'Brien Lifehouse Hospital, Camperdown, New South Wales
  - Mater Cancer Care Centre, South Brisbane, Queensland
  - Flinders Medical Center, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- France (9):
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg, Bas-Rhin
  - Institut Bergonie, Bordeaux, Gironde
  - Institut Claudius Regaud, Toulouse, Haute-Garonne
  - EDOG Institut de Cancerologie de l'Ouest, Saint-Herblain, Loire-Atlantique
  - Centre Jean Perrin, Clermont-Ferrand, Puy-de-Dôme
  - Institut Gustave Roussy, Villejuif, Val-de-Marne
  - Centre Léon Bérard Centre Régional de Lutte Contre Le Cancer, Lyon
  - CHU de Nîmes, Nîmes
  - Institute Cancer De Lorraine, Vandœuvre-lès-Nancy
- Germany (5):
  - Nationale Centrum für Tumorerkrankungen (NCT) Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Augsburg, Augsburg, Bavaria
  - Asklepios Klinik Altona, Hamburg, Hamburg
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
- Italy (9):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Istituti Fisioterapici Ospitalieri - Istituto Nazionale Tumori Regina Elena, Rome, Lazio
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Fondazione IRCCS Istituto Nazionale Dei Tumori, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Fondazione del Piemonte per l'Oncologia (IRCCS), Candiolo, Torino
  - Humanitas San Pio X, Milan
  - IRCCS - lstituto Nazionale Tumori - Fondazione G. Pascale, Napoli
- Singapore (2):
  - National University Hospital, Kent Ridge
  - National Cancer Center of Singapore, Singapore
- South Korea (5):
  - Asan Medical Center, Seoul
  - National Cancer Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul University Hospital, Seoul
  - Severance Hospital Yonsei University, Seoul
- Spain (7):
  - START MADRID_Hospital Universitario Fundacion Jimenez Diaz, Madrid, Madrid
  - START MADRID_Hospital Universitario HM Sanchinarro - CIOCC, Madrid, Madrid
  - Instituto de Investigacion Oncologica Vall d'Hebron (VHIO) - EPON, Barcelona
  - NEXT Oncology-Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - START Rioja, Rioja
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London, Middlesex
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schram AM, Fellous M, LeDuke K, Schmid A, Dumbrava EE. PYNNACLE phase II clinical trial protocol: rezatapopt (PC14586) monotherapy in advanced or metastatic solid tumors with a TP53 Y220C mutation. Future Oncol. 2025 Oct;21(24):3159-3166. doi: 10.1080/14796694.2025.2557176. Epub 2025 Sep 11. PMID 40932470
- [Derived] Papavassiliou KA, Vassiliou AG, Papavassiliou AG. Rezatapopt: A promising small-molecule "refolder" specific for TP53Y220C mutant tumors. Neoplasia. 2025 Sep;67:101201. doi: 10.1016/j.neo.2025.101201. Epub 2025 Jun 20. PMID 40543428